CLINICAL TRIAL: NCT04659499
Title: A Multicenter, Open-label, Single-arm, Phase II Clinical Trial of Nab-paclitaxel in Combination With Pyrotinib in Adjuvant Therapy for Lymph Node-negative and Small Tumor HER2-positive Breast Cancer
Brief Title: Nab-paclitaxel in Combination With Pyrotinib in Postoperative Adjuvant Therapy for HER2-positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-007
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-11

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nab-paclitaxel in combination with pyrotinib treatment group (Experimental): Nab-paclitaxel 260mg/m2 every 3 weeks for 12 weeks plus pyrotinib 240mg daily for one year
  Interventions: Drug: Nab-paclitaxel in combination with pyrotinib

INTERVENTIONS:
Drug: Nab-paclitaxel in combination with pyrotinib — Nab-paclitaxel I.V. 260mg/m2 every 3 weeks for 12 weeks plus pyrotinib oral 240mg daily for one year

SUMMARY:
This is a multicenter, open-label, single-arm, prospective, phase II study. conducted to evaluate the efficacy, safety and tolerability of nab-paclitaxel plus pyrotinib in patients with lymph node-negative and tumor size ≤3 cm, HER2 positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment subjects must have a pathological diagnosis of HER2-positive primary invasive breast cancer with an immunohistochemistry (IHC) score of 3 +, or 2 + and HER2 gene amplification by in situ hybridization (ISH) (ratio of HER2/CEP17 ≥ 2.0).
* The invasive tumor had to measure no more than 3cm and with histologically confirmed lymph node-negative or one lymph node micrometastasis (T ≤ 3 cm, N0/N1mi, M0).
* Tumor should has known ER/PR hormone receptor status.
* All patients must be women above18 years old with Eastern Cooperative Oncology Group score 0 to 1.
* Adequate hematopoietic function and organ function as defined as follows: neutrophil count ≥ 1.5 x 109/L; Platelet count ≥ 90 × 109/L; Hemoglobin ≥ 90 g/L; total bilirubin ≤ 1.5 × ULN; alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 3 × ULN; serum creatinine Cr ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula).
* left ventricular ejection fraction (LVEF) ≥ 50% and Electrocardiogram Fridericia-corrected QT interval (QTcF) ≤ 480 ms.
* Provide written informed consent.

Exclusion Criteria:

* Clinical or radiologic evidence of local or regional recurrence of disease or metastatic disease prior to or at the time of study entry.
* Previous treatment with chemotherapeutic drugs, or tyrosine kinase inhibitors targeting HER2 (lapatinib, neratinib or pyrotinib, etc.).
* Other malignancies within the past 5 years, excluding cured cervical carcinoma in situ, cutaneous basal cell carcinoma, or cutaneous squamous cell carcinoma.
* Inability to swallow, chronic diarrhea, or intestinal obstruction.
* Known to be allergic to the drug components.
* Have a history of immunodeficiency, including HIV positive, HCV positive, active viral hepatitis B or other immunodeficiency diseases.
* Have a history of organ transplantation.
* Pregnant, lactating female patients, or female patients who are unwilling to take effective contraceptive.
* Any heart disease, including: (1) arrhythmia; (2) myocardial infarction; (3) heart failure.
* Any other concomitant diseases assessed by investigator as unsuitable for study.
* Previous history of definite neurological or psychiatric disorders.
* Concomitant use of CYP3A4 inhibitors or inducers or drugs that prolong the QT interval.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
3-year-DFS | From the start of treatment to 3 years
  3-years-disease free survival rate

SECONDARY OUTCOMES:
AEs+SAEs | from the first drug administration to within 28 days for the last pyrotinib dose
  Adverse Events and Serious Adverse Events are described in terms of CTC AE 5.0

REFERENCES:
- [Derived] Wang C, Zhou Y, Lin Y, Mao F, Guan J, Zhang X, Shen S, Wang X, Zhang Y, Pan B, Zhong Y, Peng L, Cao X, Yao R, Zhou X, Xu C, Xu Y, Sun Q. Rationale and design of a phase II trial of pyrotinib in combination with nab-paclitaxel as adjuvant therapy for N0/N1mi, HER2 + early breast cancer (PHAEDRA). BMC Cancer. 2022 Mar 14;22(1):269. doi: 10.1186/s12885-022-09346-1. PMID 35287613